CLINICAL TRIAL: NCT01764204
Title: Intensive Hospital-based Adverse Drug Reaction Monitoring Study On Patients Treated By Qingkailing Injection In The Next Two Years
Brief Title: Hospital Intensive Monitoring of Adverse Drug Reactions of Qingkailing Injection In The Next Two Years
Status: Completed | Type: Observational
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Other Study IDs: Qingkailing-V5.0
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Adverse Drug Events; Adverse Drug Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Qingkailing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood of the patient with severe adverse drug reactions
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Qingkailing Injection
  Interventions: Drug: Qingkailing Injection

INTERVENTIONS:
Drug: Qingkailing Injection — Qingkailing Injection is a kind of natural product injection made from Chinese herbs, which has been used to treat cerebral ischemia for decades in China. The main bioactive ingredients of this injection include Baicalin, Jasminoidin, Ursodeoxycholic Acid, Concha Margaritifera,etc.
  Other Names: Shineway Qingkailing Injection

SUMMARY:
To highlight the incidence of adverse reactions of Qingkailing Injection.

ELIGIBILITY:
Inclusion Criteria:

* all the patients treated by Qingkailing Injection in the certain centers(hospitals) in the next 2 years.
* in accordance with ethics requirements.

Exclusion Criteria:

* none.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all the patients treated by Qingkailing Injection in the certain centers(hospitals) in the next 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 30840 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
incidence of severe adverse drug reactions | 2 years

SECONDARY OUTCOMES:
incidence of adverse drug reactions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Ph.D., M.D., Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences
Locations (48):
- China (48):
  - National Defense University Hospital of People's Liberation Army, Beijing, Beijing Municipality
  - Ren'ai Hospital, Shenzhen, Guangdong
  - Chinese Medicine Hospital of Deqing County, Zhaoqing, Guangdong
  - Chinese Medicine Hospital of Gaoyang County, Baoding, Hebei
  - Gaoyang County Hospital, Baoding, Hebei
  - The Third People's Hospital of Xiong County, Baoding, Hebei
  - Chinese Medicine Hospital of Xiong County, Baoding, Hebei
  - Chinese Medicine Hospital of Tang County, Baoding, Hebei
  - People's Hospital of Tang County, Baoding, Hebei
  - Chinese Medicine Hospital of Handan City, Handan, Hebei
  - The First Hospital of Yongnian District, Handan, Hebei
  - The Second Hospital of Yongnian District, Handan, Hebei
  - Central Hospital of Shijiazhuang City, Shijiazhuang, Hebei
  - Hebei Chest Hospital, Shijiazhuang, Hebei
  - Chinese Medicine Hospital of Shijiazhuang City, Shijiazhuang, Hebei
  - Central Hospital of Qinghe County, Xingtai, Hebei
  - Chinese Medicine Hospital of Xingtai City, Xingtai, Hebei
  - Eye Hospital of Xingtai City, Xingtai, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Chinese Medicine Hospital of Qinghe County, Xingtai, Hebei
  - The Second Hospital of Bayan County, Harbin, Heilongjiang
  - Luohe Hospital of Chinese Medicine, Luohe, Henan
  - Central Hospital of Sanmenxia City, Sanmenxia, Henan
  - People's Hospital of Shan County, Sanmenxia, Henan
  - The First People's Hospital of Lingbao, Sanmenxia, Henan
  - Chinese Medicine Hospital of Xinxiang City, Xinxiang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - People's Hospital of Yanjin County, Xinxiang, Henan
  - Chinese Medicine Hospital of Fengqiu County, Xinxiang, Henan
  - People's Hospital of Fengqiu County, Xinxiang, Henan
  - People's Hospital of Yuanyang County, Xinxiang, Henan
  - People's Hospital of Xinzheng City, Xinzheng, Henan
  - Third Affiliated Hospital of Henan College of Traditional Chinese Medicine, Zhengzhou, Henan
  - Chinese Medicine Hospital of Xinzheng, Zhengzhou, Henan
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Central Hospital of Liaocheng City, Liaocheng, Shandong
  - Veterans'Hospital, Liaocheng, Shandong
  - Chinese Medicine Hospital of Dongchangfu District, Liaocheng, Shandong
  - Chinese Medicine Hospital of Chiping County, Liaocheng, Shandong
  - YangGuXian People's Hospital, Liaocheng, Shandong
  - Chinese Medicine Hospital of Linqing, Liaocheng, Shandong
  - Chinese Medicine Hospital of Gaotang County, Liaocheng, Shandong
  - Community Health Center of Duqiao, Weinan, Shanxi
  - Chinese Medicine Hospital of Sanyuan County, Xianyang, Shanxi
  - People's Hospital of Fuyuan County, Qujing, Yunnan
  - Chinese Medicine Hospital of Luliang County, Qujing, Yunnan
  - People's Hospital of Luliang County, Qujing, Yunnan
  - Chinse Medical Hospital of Shizong County, Qujing, Yunnan

REFERENCES:
- [Derived] Yao Q, Wei T, Qiu H, Cai Y, Yuan L, Liu X, Li X. Epigenetic Effects of Natural Products in Inflammatory Diseases: Recent Findings. Phytother Res. 2025 Jan;39(1):90-137. doi: 10.1002/ptr.8364. Epub 2024 Nov 8. PMID 39513382